CLINICAL TRIAL: NCT04789382
Title: Clinical Biocompatibility of Three Daily Wear Monthly Replacement Silicone Hydrogel Contact Lenses With Two Multi-purpose Disinfecting Solution Combinations
Brief Title: Three Daily Wear Monthly Replacement Silicone Hydrogel Contact Lenses With Two Multi-purpose Disinfecting Solution Combinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-E007
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Refractive Errors
Keywords: contact lens; contact lens solution
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sequence 1 (Other): LID018869+RepleniSH in the right eye and Biofinity+RepleniSH in the left eye (first wear period), followed by PV+Biotrue in the right eye and LID018869+Biotrue in the left eye (second wear period). Each wear period will be 2 hours.
  Interventions: Device: LID018869+RepleniSH; Device: LID018869+Biotrue; Device: Biofinity+RepleniSH; Device: PV+Biotrue
- Sequence 2 (Other): Biofinity+RepleniSH in the right eye and LID018869+RepleniSH in the left eye (first wear period), followed by LID018869+Biotrue in the right eye and PV+Biotrue in the left eye (second wear period). Each wear period will be 2 hours.
  Interventions: Device: LID018869+RepleniSH; Device: LID018869+Biotrue; Device: Biofinity+RepleniSH; Device: PV+Biotrue
- Sequence 3 (Other): LID018869+Biotrue in the right eye and PV+Biotrue in the left eye (first wear period), followed by Biofinity+RepleniSH in the right eye and LID018869+RepleniSH in the left eye (second wear period). Each wear period will be 2 hours.
  Interventions: Device: LID018869+RepleniSH; Device: LID018869+Biotrue; Device: Biofinity+RepleniSH; Device: PV+Biotrue
- Sequence 4 (Other): PV+Biotrue in the right eye and LID018869+Biotrue in the left eye (first wear period), followed by LID018869+RepleniSH in the right eye and Biofinity+RepleniSH the left eye (second wear period). Each wear period will be 2 hours.
  Interventions: Device: LID018869+RepleniSH; Device: LID018869+Biotrue; Device: Biofinity+RepleniSH; Device: PV+Biotrue

INTERVENTIONS:
Device: LID018869+RepleniSH — Lehfilcon A silicone hydrogel spherical contact lens pre-cycled (pre-soaked prior to dispense) with OPTI-FREE® RepleniSH® multi-purpose disinfecting solution (RepleniSH)
Device: LID018869+Biotrue — Lehfilcon A silicone hydrogel spherical contact lens pre-cycled (pre-soaked prior to dispense) with Biotrue® multi-purpose solution (Biotrue)
Device: Biofinity+RepleniSH — Comfilcon A silicone hydrogel spherical contact lens pre-cycled (pre-soaked prior to dispense) with OPTI-FREE® RepleniSH® multi-purpose disinfecting solution (RepleniSH)
Device: PV+Biotrue — Balafilcon A silicone hydrogel spherical contact lens pre-cycled (pre-soaked prior to dispense) with Biotrue® multi-purpose solution (Biotrue)

SUMMARY:
The purpose of this study is to evaluate corneal staining observed after 2 hours of wear with an investigational contact lens against both PureVision contact lenses pre-cycled with Biotrue and Biofinity contact lenses pre-cycled with RepleniSH.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1:1:1 manner to receive one of 4 regimen sequences with lens and multipurpose disinfection solution (MPDS) combinations. The expected duration of subject participation in the study is approximately 1 week with 2 study visit days.

ELIGIBILITY:
Key Inclusion Criteria:

* Understand and sign an Informed Consent;
* Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Manifest cylinder of less than or equal to 1.50 diopter (D) in each eye;
* Best corrected visual acuity (BCVA) better than or equal to 20/25 Snellen in each eye;
* Willing to stop wearing habitual contact lenses for the duration of study lens exposure and during the washout period.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any eye condition or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* Eye surgery, as specified in the protocol;
* Dry eye; use of artificial tears, as specified in the protocol;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Alcon Investigator 6565, Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one investigative site located in the United States.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Groups:
- Sequence 1: LID018869+RepleniSH in the right eye and Biofinity+RepleniSH in the left eye (first wear period), followed by PV+Biotrue in the right eye and LID018869+Biotrue in the left eye (second wear period). Each wear period was 2 hours.
- Sequence 2: Biofinity+RepleniSH in the right eye and LID018869+RepleniSH in the left eye (first wear period), followed by LID018869+Biotrue in the right eye and PV+Biotrue in the left eye (second wear period). Each wear period was be 2 hours.
- Sequence 3: LID018869+Biotrue in the right eye and PV+Biotrue in the left eye (first wear period), followed by Biofinity+RepleniSH in the right eye and LID018869+RepleniSH in the left eye (second wear period). Each wear period was 2 hours.
- Sequence 4: PV+Biotrue in the right eye and LID018869+Biotrue in the left eye (first wear period), followed by LID018869+RepleniSH in the right eye and Biofinity+RepleniSH the left eye (second wear period). Each wear period was 2 hours.
Period: First Wear Period (2 Hours)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout (Day of & Day Prior to Visit 3)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Second Wear Period (2 Hours)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lens, whether or not presoaked in the study multi-purpose disinfecting solution (MPDS)
Groups:
- Sequence 2: Biofinity+RepleniSH in the right eye and LID018869+RepleniSH in the left eye (first wear period), followed by LID018869+Biotrue in the right eye and PV+Biotrue in the left eye (second wear period). Each wear period was 2 hours.
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (5.4) | 29.0 (5.9) | 36.0 (6.8) | 31.6 (6.3) | 31.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 8 | 27
  Male | 3 | 2 | 3 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 8 | 8 | 7 | 9 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 9 | 9 | 8 | 9 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Area of Corneal Staining
Description: A slit lamp examination was performed by the investigator to assess corneal staining. Percent of solution-related corneal staining area was assessed first in each of the 5 corneal regions: central, superior, nasal, inferior, and temporal. The average of corneal staining area was then calculated as the average over all 5 regions. Each eye was treated differently and was graded separately. No hypotheses were formulated; no inferences were made, and only descriptive statistics were used in the reporting.
Time Frame: Hour 2 (each wear period)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of area
Units Other Than Participants: eyes
Groups:
- LID018869+RepleniSH: LID018869+RepleniSH worn for 2 hours in the right eye or left eye and during Period 1 or Period 2, as randomized
- Biofinity+RepleniSH: Biofinity+RepleniSH worn for 2 hours in the right eye or left eye and during Period 1 or Period 2, as randomized
- LID018869+Biotrue: LID018869+Biotrue worn for 2 hours in the right eye or left eye and during Period 1 or Period 2, as randomized
- PV+Biotrue: PV+Biotrue worn for 2 hours in the right eye or left eye and during Period 1 or Period 2, as randomized
Arm/Group | LID018869+RepleniSH | Biofinity+RepleniSH | LID018869+Biotrue | PV+Biotrue
Number analyzed (Participants) | 36 | 36 | 36 | 36
Number analyzed (eyes) | 36 | 36 | 36 | 36
percentage of area | 2.93 (8.86) | 0.45 (1.03) | 6.06 (14.75) | 3.52 (11.87)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 1 week.
Description: An AE was defined at any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the test article. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. At Risk" population of pretreatment and non-ocular AEs is reported in units of subjects; all other AE populations are reported in units of eyes.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID018869+RepleniSH Ocular; Biofinity+RepleniSH Ocular; LID018869+Biotrue Ocular; PV+Biotrue Ocular: Events reported in this group occurred while exposed to the study contact lenses
- All Nonocular: Events reported in this group occurred while left and right eyes were exposed to different study lenses as per randomized regimen sequence
Arm/Group | Pretreatment | LID018869+RepleniSH Ocular | Biofinity+RepleniSH Ocular | LID018869+Biotrue Ocular | PV+Biotrue Ocular | All Nonocular
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT04789382/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT04789382/SAP_001.pdf